CLINICAL TRIAL: NCT06840912
Title: Electroencephalographic Biofeedback Therapy in Heroin Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa El sayed Ali Elhout, Resident of Neuropsychiatry, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS20/1/23
Record Dates: First submitted 2025-02-12; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Electroencephalographic; Biofeedback Therapy; Heroin; Craving
MeSH Terms: interventions — Biofeedback, Psychology; Drug Therapy; Control Groups

STUDY DESIGN:
Intervention Model Description: we use EEG Biofeedback device for correction of abnormal wave amplitude in heroin addict patients after three months of abstinence aiming to decrease craving beside traditional pharmacotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EEG biofeedback beside pharmacotherapy group (Experimental): Patients with heroin use disorder diagnosed according to DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders 5th edition), treated by pharmacological ( symptomatic treatment only ) in addition to electroencephalographic (EEG) biofeedback device after 3 months of abstinence.
  Interventions: Other: Pharmacological in addition to electroencephalographic (EEG) biofeedback
- pharmacotherapy group (Other): Patients with heroin use disorder taken as control group matching with patients group in terms of age, gender, daily heroin use and duration of use , treated only by pharmacotherapy ( symptomatic treatment only).
  Interventions: Drug: Pharmacotherapy

INTERVENTIONS:
Other: Pharmacological in addition to electroencephalographic (EEG) biofeedback — Patients with heroin use disorder diagnosed according to DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders 5th edition), treated by pharmacological in addition to electroencephalography (EEG) biofeedback after 3 months of abstinence.
  Arms: EEG biofeedback beside pharmacotherapy group
Drug: Pharmacotherapy — Patients with heroin use disorder taken as control group matching with patients group treated only by pharmacotherapy
  Other Names: Control group
  Arms: pharmacotherapy group

SUMMARY:
The aim of this work is to assess the effectiveness of electroencephalography (EEG) biofeedback in management of heroin craving .

DETAILED DESCRIPTION:
Substance use disorder is characterized by physiological dependence accompanied by the withdrawal syndrome upon abstinence from the drug, psychological dependence, tolerance, expressed in the escalation of the dose needed to achieve a desired euphoric state , and craving which is a pathological motivational state that leads to active drug-seeking behavior which leads to relapse . substance use disorder is a chronic, relapsing mental disease that results from the prolonged effects of drugs on the brain.

Narcotic drugs addiction is recurrent and chronic mental illness with severe motivational disorders and loss of behavioral control.

Craving is a penchant and persistent desire of drugs consumption, if it is not met, will have Psychological and physical sufferings, such as fatigue, anorexia, anxiety, insomnia, aggression, and depression. Also, voracity is very strong sense and urgent desiring to one thing, so that any possibility of focusing on something other than the asked subject is impossible. EEG biofeedback is an operant conditioning technique used to reinforce certain waves and inhibit others, in heroin patients, there is a decrease in mean alpha wave and SMR wave amplitude which persist and excess beta wave activity which abolished after 3 months of abstinence , increase in mean SMR wave amplitude lead to decrease impulsivity and improve attention , increase in alpha wave mean amplitude , decrease anxiety which accompany craving .

ELIGIBILITY:
Inclusion Criteria:

* All persons included in this study are males.
* Persons aged from 20 to 50 years.
* Addicts abusing one substance only (heroin).
* They had received at least 3 months of pharmacological treatment.
* complete blood and urine test had been taken from all participants.
* Subjects must be able to comprehend and perform study related information and tasks , are willing to complete study procedures.

Exclusion Criteria:

* Addicts abusing other substances with heroin.
* History of any neurological disorder that would result in abnormal electroencephalography (EEG) activity such as seizure disorders, stroke.
* Currently on a medication which is known to alter electroencephalography (EEG) activity as anticonvulsant, anticholinergic or benzodiazepine.
* Age younger than 20 and older than 50 years.
* Patients suffering from any psychiatric disorders in addition to heroin abuse.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All persons included in this study are males.
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Brief substance craving scale( BSCS) | 14 months
  Brief substance craving scale ( BSCS): It is a self-report instrument to assess craving for heroin abuse over a 24 hour period. Patients were asked to complete a scale, rating the intensity, frequency and length of their cravings. Ratings were then scored on a scale of 0 to 12 (0) meaning no cravings- (12) meaning the patient was experiencing severe craving.
  1. The intensity of my craving, that is, how much I desired this drug in the past 24 hours was:
     a- None at all. b- Slight. c-Moderate. d- Considerable. e- Extreme
  2. The frequency of my craving, that is, how often I desired this drug in the past 24 hours was:
     a- Never b- Almost never. c-Several times. d- Regular. Performed at baseline to both groups before starting EEG Biofeedback . At the next day after completion of twenty sessions of EEG Biofeedback. After 1 month follow up. After 2 month follow up. There was a decrease in brief substance craving scale in experimental group in comparison to control group.

SECONDARY OUTCOMES:
Electroencephalographic (EEG) biofeedback | 14 months
  Assessment of mean brain waves amplitude by EEG biofeedback device "Thought technology Ltd Flex Comp Infinti" ( used as treatment and assessment device ) , only assessment methods for both group, and treatment method to experimental group.
  we use two protocols in experimental group : ten sessions of SMR /Theta protocol and another ten of alpha / Theta protocol every other day for 50 minutes we asses mean SMR wave amplitude to both groups at base line , then after completion of sessions , one and two months after.
  we assess also mean Alpha wave amplitude to both groups at base line , then after completion of sessions , one and two months after.
  there was an increase in both SMR and Alpha wave mean amplitude in experimental group in comparison to control group, this means decrease impulsivity and increase attention (SMR wave amplitude increase ), decrease anxiety by increase in mean alpha wave amplitude .
General Health Questionnaire (GHQ-12) | 14 months
  The 12-Item General Health Questionnaire (GHQ-12) consists of 12 items, each one assessing the severity of a mental problem over the past few weeks using a 4-point Likert-type scale (from 0 to 3). The score was used to generate a total score ranging from 0 to 36. The positive items were corrected from 0 (always) to 3 (never) and the negative ones from 3 (always) to 0 (never). High scores indicate worse health. It includes three factors, namely Anxiety and Depression, Social Dysfunction, and Loss of Confidence.
  1. Score from (0-15): normal without distress.
  2. Score from (16-25): mild distress.
  3. Score more than or equal 25: severe distress.
     * It was preformed at baseline before starting EEG Biofeedback.
     * At the next day after completion of twenty sessions of EEG Biofeedback to experimental group I , and assessment of control group at the same time.
     * After 1 month follow up.
     * After 2 month follow up. it decreased in experimental group in comparison to control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author